CLINICAL TRIAL: NCT07014163
Title: Evaluating the Efficacy and Safety of Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.) Injection in the Management of Superficial Lipomas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Espad Pharmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMB.ESP.KB.IV.03
Record Dates: First submitted 2025-05-20; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Lipoma
MeSH Terms: conditions — Lipoma

STUDY DESIGN:
Intervention Model Description: before/after clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Embella (Deoxycholic acid, produced by Espad Pharmed Co.) (Experimental): During each treatment, 0.1 mL or 0.15 mL of a 10 mg/mL deoxycholic acid solution will be injected into every 1*1 cm2 of the lipoma using an insulin syringe with a 1cm needle attached (the max volume of injection is 2 cc in each treatment session). Pressure will be applied directly to the site of injection for several seconds to prevent local bleeding and an adhesive dressing will be applied.
  The injection will be done at visit 1 (day 0) for everyone and at visits 2 (week 4) and 3 (week 8) as touch-up injections if needed (treatment will be continued until the patient is satisfied with the lipoma's response to the injection, for a max of 3 injections).
  Interventions: Device: Embella (Deoxycholic acid, produced by Espad Pharmed Co.)

INTERVENTIONS:
Device: Embella (Deoxycholic acid, produced by Espad Pharmed Co.) — 0.1 mL or 0.15 mL of a 10 mg/mL deoxycholic acid solution will be injected into every 1*1 cm2 of the lipoma using an insulin syringe with a 1cm needle attached (the max volume of injection is 2 cc in each treatment session).

SUMMARY:
Lipoma is a relatively common, slow-growing mesenchymal neoplasm originating from adipose tissue. Patients seek treatment for lipomas for various reasons, such as concerns about their growth and spread, aesthetic issues, or worries about the compressive effects of the lipoma. Lipomas are typically removed surgically through excision, which can have complications including bleeding, infection, scarring, and recurrence. Other mentioned treatment methods include liposuction, laser, and medicinal approaches.

Purified synthetic deoxycholic acid has been introduced as the first pharmacological intervention approved by the FDA for the reduction of submental fat. Deoxycholic acid is a type of bile acid that, due to its ability to cause non-selective cell lysis and disruption of adipocyte membranes (adipocytolysis), leads to emulsification of fat in the intestine.

This is an interventional (pre-post), single-arm, and open-label study to evaluate the efficacy and safety of Embella (Deoxycholic acid, produced by Espad Pharmed Co.) for the management of superficial lipomas.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aging between 18 to 65 years
2. Having at least one lipoma (based on clinical and sonographic diagnosis), which is accessible for treatment and assessment and is quantifiable along at least 2 perpendicular diameters and lower than 2 centimeter in depth, with the following characteristics:

   * History of slow growth followed by dormancy
   * Being stable for at least 6 months
   * Greatest length by greatest perpendicular width between 4 and 4 square centimeters
   * Inclusive discrete, oval to rounded in shape, not hard or attached to underlying tissue
   * Located on the trunk, upper and lower limbs, far from main and vulnerable neurovascular structures
3. Stable body weight with a body mass index of less than 30 kg/m² in the past three months
4. Signed informed consent
5. Ability to follow study instructions and likely to complete all required visits
6. Agreement to abstain from any treatment for lipomas during the study

Exclusion Criteria:

1. Any medical and physical conditions (for example, high blood pressure or respiratory, cardiovascular, liver, neurological, or thyroid disorders) that, in the opinion of the attending physician, affect the evaluation of the efficacy and safety of the product.
2. Known allergy or sensitivity to the study medication or its components
3. Females who are pregnant or breastfeeding, or expecting to conceive children within the projected duration of study
4. Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study and for the duration of the study.
5. Previous treatment for lipomas
6. Subjects planning a surgical procedure for lipoma during the study or at any time that may affect the evaluation
7. Subjects with volume deficit due to trauma, abnormalities in adipose tissue related to immune-mediated diseases such as generalized lipodystrophy (e.g., juvenile dermatomyositis), partial lipodystrophy (e.g., Barraquer-Simons syndrome) or HIV-related disease
8. Evidence of recent alcohol or drug abuse
9. Medical and/or psychiatric problems that are severe enough to interfere with the study results
10. Known bleeding disorder or receiving medication that will likely increase the risk of bleeding after injection
11. Having a tendency to develop hypertrophic scarring
12. Having a history of anaphylaxis or allergy to lidocaine (or any amide-based anesthetics), hyaluronic acid products, or Streptococcal protein
13. Having an active inflammation, dermatoses, infection, cancerous or precancerous lesion, or unhealed wound in the site of lipoma
14. Having a condition or being in a situation that, in the investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of calculated volume change of lipoma in participants | Baseline and week 16
  Percentage of calculated volume change from baseline to week 16 based on ultrasound evaluation in participants
Percentage of lipoma size change in participants | Baseline and week 16
  Percentage of lipoma size change from baseline to week 16 based on both ultrasound evaluation and objective evaluation (using flexible meter) in participants
Percentage of participant with lipoma size change more than 50% | Baseline and week 16
  Percentage of participant with size change more than 50% from baseline to week 16
Score of patient satisfaction | Week 16
  The score is evaluated by the answers of two questions:
  1. How satisfied are you with the result of your injections? The scales are from 1 to 5, 1 indicating very dissatisfied, and 5 indicating very satisfied.
  2. Knowing what you know now, how likely is it that you would choose this method again for your initial problem? The scales are: 1 indicating very likely, 3 indicating somewhat likely, and 5 indicating unlikely.

SECONDARY OUTCOMES:
Percentage of participants requiring touch-up injection | Week 4 and week 8
  Percentage of participants requiring touch-up injection (week 4 and week 8)
Percentage of participants requiring surgical removal | Week 16
  Percentage of participants requiring surgical removal in 4 months after injections
Number of injections needed to achieve favorable result | Week 16
  Number of injections needed to achieve favorable result
The change in diameter of lipoma compared to baseline | Baseline, week 4, and week 8
  The change in diameter of lipoma compared to baseline (week 4 and 8) based on ultrasound evaluation
The change in volume of lipoma compared to baseline | Baseline, week 4, and week 8
  The change in volume of lipoma compared to baseline (week 4 and 8) based on ultrasound evaluation
The change in depth of lipoma compared to baseline | Baseline, week 4, and week 8
  The change in depth of lipoma compared to baseline (week 4 and 8) based on ultrasound evaluation
Safety assessment by evaluation of the severity of adverse events (AEs) | Screening visit, Visit 1 (Day 0), Visit 2 (week 4), Visit 3 (week 8), Visit 4 (week 16)
  The severity of AEs is assessed at all visits, based on the physician's judgment.
Safety assessment by evaluation of the seriousness of adverse events (AEs) | Screening visit, Visit 1 (Day 0), Visit 2 (week 4), Visit 3 (week 8), Visit 4 (week 16)
  The seriousness of AEs is assessed at all visits, in accordance with the International Council for Harmonization (ICH-E2B) guidelines.
Safety assessment by evaluation of causality of adverse events (AEs) | Screening visit, Visit 1 (Day 0), Visit 2 (week 4), Visit 3 (week 8), Visit 4 (week 16)
  The causality of AEs is assessed at all visits, based on World Health Organization (WHO) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Balighi, Principal Investigator — Department of Dermatology, Razi Hospital, Tehran University of Medical Sciences, Tehran, Iran.
Locations (2):
- Iran (2):
  - Orchid Pharmed, Medical Department, Tehran, Tehran Province
  - Razi hospital, Tehran

IPD SHARING:
Plan to Share IPD: No
Data produced in the present study are available upon reasonable request from the investigators.